CLINICAL TRIAL: NCT01736007
Title: Childhood Alopecia Areata Study: Part 1: Feasibility of the 308-nm Excimer Laser in Treatment of Patch Type Alopecia Areata in Pediatric Patients
Brief Title: Childhood Alopecia Areata Study Using the 308-nm Excimer Laser
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: was not able to recruit participants
Sponsor: Phoenix Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PCH-derm001; IDE Number: G110232/S2 (Other: FDA)
Record Dates: First submitted 2012-11-01; First posted 2012-11-28 (Estimated); Last update posted 2014-10-31 (Estimated); Status verified 2014-10

CONDITIONS: Alopecia Areata
Keywords: alopecia areata child; scalp
MeSH Terms: conditions — Alopecia Areata

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Liquid light guide tip on laser (Sham Comparator): Excimer laser treatment with 308-nm excimer laser with guide tip applied to alopecia patch twice a week.
  Interventions: Device: Liquid light guide tip on laser
- 308-nm excimer laser to alopecia patch (Active Comparator): Laser treatment with 308-nm excimer laser procedure to alopecia patch twice a week with increasing fluence as tolerated.
  Interventions: Device: 308-nm excimer laser to alopecia patch

INTERVENTIONS:
Device: 308-nm excimer laser to alopecia patch — MED dosing as per protocol with beginning at 50 mJ/cm2 below MED with increases by 50mJ/cm2 every 2 treatments as tolerated. Maximum dosing would be 850mJ.Treatments given twice a week for 12 weeks.
  Other Names: PhotoMedex XTRAC XL Excimer Laser System, Model AL 8000
  Arms: 308-nm excimer laser to alopecia patch
Device: Liquid light guide tip on laser — Sham treatment involves placement of liquid light guide tip developed by the laser company which attaches to the end of the hand wand and blocks the laser light from passing to the target. Patients are treated twice a week for 12 weeks.
  Other Names: Liquid light guide tip applied to Excimer laser
  Arms: Liquid light guide tip on laser

SUMMARY:
Alopecia Areata (AA) is a skin restricted autoimmune disease of the hair follicle, resulting in hair loss of the scalp, and in severe cases of the entire body. AA is the second most common cause of alopecia in childhood; no FDA-approved treatments exist. The use of focused narrow-band ultraviolet-B light via the excimer laser is a common treatment for many skin diseases in patients of all ages. In this study, the feasibility of the 308-nm excimer laser for treatment of patch type AA of the scalp will be examined. We anticipate the excimer laser will be safe and a feasible option for patients with patch type AA. The excimer laser may represent a novel treatment for childhood AA and no comparison or large studies currently exist in the literature.

Hypotheses The 308-nm excimer laser procedure is a feasible, well-tolerated and safe treatment for patch type alopecia areata of the scalp in children.

DETAILED DESCRIPTION:
The goal of this study is to assess the feasibility, safety and response to treatment of the use of the 308-nm excimer laser in children (age 6-17 years) diagnosed with patch type alopecia areata involving the scalp, present for more than 6 months duration. Patients meeting the inclusion criteria will be randomly enrolled in a treatment group or placebo group. Response to treatment during and after the 12-week laser treatment course will be measured in terms of hair regrowth utilizing the SALT score and 2 blinded evaluations of subject photographs.

Specific Aims Evaluate the feasibility and safety of twice-weekly excimer laser treatments over a period of 12 weeks. Measures will include side effects, response to treatment (hair growth), tolerability of therapy, attrition, attendance, and overall satisfaction with this treatment modality.

ELIGIBILITY:
Inclusion Criteria:

1. Children 6-17 years old, diagnosed with patch type alopecia areata for a minimum of 6 months prior to enrollment involving the scalp.
2. A Parent/guardian consent and child assent (in those 8 years old or greater) must be obtained.
3. Parent/guardian and patient agree to MED dose test with a 24 hour follow up visit and a 12 week period of twice weekly treatment in either group, as well as baseline, interim and end of study visits.
4. Parent/guardian and child must be able to understand English or Spanish to participate.
5. Parent/guardian must agree to have the patient undergo a washout period of 6 weeks prior to the enrollment of the study if the patient is currently on treatment of any kind (oral and/or topical) for AA.

Exclusion Criteria:

1. Children who have been diagnosed with an autoimmune skin disease or photosensitivity disorder.
2. Children who have been using topical steroids to the scalp, have other scalp disease or are using injected or oral steroids, biologic agents or chemotherapy for other medical conditions.
3. Children under current treatment for other skin conditions with oral medications (such as an oral corticosteroid) and/or topical treatments such as topical corticosteroids that may affect hair regrowth. Specifically, for topical medications, any child that requires the use of class 1-2 topical corticosteroids will be excluded.

3. Any subject who is currently experiencing significant spontaneous regrowth of terminal hair.

4. Patients with alopecia universalis, totalis, ophiasis pattern or diffuse AA may not participate in this feasibility study.

4. Parent/guardian who do not consent or children who do not assent to participate.

5. Any subject who has had AA for less than 6 months and is not willing to undergo a 6 week wash-out period prior to start of the study.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2012-08; Primary Completion 2013-06 (Estimated); Study Completion 2014-08 (Estimated)

PRIMARY OUTCOMES:
The goal of this study is to assess the feasibility, safety and response to treatment of the use of the 308-nm excimer laser in children diagnosed with patch type alopecia areata involving the scalp, present for more than 6 months duration | 9 months
  Response to treatment during and after the 12-week laser treatment course will be measured in terms of hair regrowth utilizing the SALT score and 2 blinded evaluations of subject photographs. Follow up post treatment at 36 weeks and 48 weeks.

SECONDARY OUTCOMES:
Evaluate the feasibility and safety of twice-weekly excimer laser treatments over a period of 12 weeks | 48 weeks
  Measures will include side effects, response to treatment (hair growth), tolerability of therapy, attrition, attendance, and overall satisfaction with this treatment modality.

CONTACTS AND LOCATIONS:
Overall Officials: Harper N Price, MD, Principal Investigator — Phoenix Children's Hospital; Judith AJ O'Haver, PhD, Principal Investigator — Phoenix Children's Hospital
Locations (1):
- Phoenix Children's Hospital, Phoenix, Arizona, United States